CLINICAL TRIAL: NCT03567226
Title: Leveraging WeChat Social-Media and Messaging Platform to Increase Physical Activity in Chinese Glaucoma Patients: A Pilot Study
Brief Title: Leveraging WeChat Social-Media and Messaging Platform to Increase Physical Activity in Chinese Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00172315
Record Dates: First submitted 2018-05-29; First posted 2018-06-25 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Counseling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will be enrolled into a WeChat Group to receive reminders to exercise and health education materials.
  Interventions: Behavioral: WeChat Group
- Control Group (Active Comparator): Controls will receive a handout telling them to increase walking and that walking may be helpful for the eye at the return visit.
  Interventions: Behavioral: Counselling

INTERVENTIONS:
Behavioral: WeChat Group — Consenting participants will be randomized to either the intervention or the control arm after successfully wearing an accelerometer for one week. The WeChat Group will be a community forum to share information, encourage each other, and receive communications from the study team. In addition, the study team will disseminate the following information through the group:
  1. Daily/Weekly Reminders to exercise
  2. Health education materials regarding glaucoma and general health and exercise
  3. Motivational content
  4. Surveys to gauge what information participants found most interesting and useful to help them exercise
  Arms: Intervention Group
Behavioral: Counselling — Study participants in the control group will receive a handout telling them to increase walking and will be counseled that walking may be helpful for the eye at the return visit
  Arms: Control Group

SUMMARY:
The positive effects of exercise on ocular health are known, but modern lifestyles have made it difficult to incorporate physical activity into the daily lives of the Chinese population. Recent studies suggest that exercise plays an important role in lowering intraocular pressure (IOP) by protecting retinal ganglion cells (RGCs) in glaucoma patients as well as other potential neuroprotective benefits. Increasing the amount of physical activity within the Chinese glaucoma population may have marked effects on health outcomes and coincides with the Chinese government's efforts to make exercise an urgent public health priority. There is a need for innovative, cost-effective, and proven interventions to promote exercise behavior change and social media platforms may be able to fill this niche. WeChat is China's largest and most frequently used social media and messaging application with an estimated 570 million users. The platform has been found to be a useful tool in healthcare settings to promote weight-loss, health literacy, and patient adherence in Chinese populations. This study is a 5-weeks randomized control trial with three total study visits. 80 patients from an academic glaucoma clinic in Wenzhou Medical College will be randomized into two groups. The intervention group will be enrolled into an Official WeChat Group and receive periodic reminders to exercise, health education materials, and motivational incentives. The control group will receive weekly reminders and leaflets at the first clinic visit. Patients' daily step data will be monitored using an Accelerometer WGT3X-BT. The intervention duration will include an initial clinic visit, a one-week follow-up after wearing the accelerometer, and then a subsequent one-month follow-up visit after wearing the accelerometer. At the one-week visit the patient will be randomized and at the subsequent one-month visit there will be a close-out discussion about the study. In addition to collecting step data at clinic visits, investigators will also measure patients' visual field tests, optical coherence tomography angiography (angio-OCT), and intraocular pressure (IOP) using Goldmann Tonometry. The investigators' hypothesis is that using an Official WeChat Patient Group will be a robust and effective stimulus to increase physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma diagnosis
* Age 40 years and above
* Ability to sign informed consent
* Ability to use WeChat

Exclusion Criteria:

* Patients with severe heart, lung, or kidney disease which may prevent them from exercising
* Patients who self-report walking 12,000 steps or more per day

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Efficacy of using WeChat as an intervention to increase physical activity in Chinese glaucoma patients | 5 weeks
  The primary outcome variable will be the number of daily steps taken over the course of one month for each participant. This outcome will be measured by having participants wear the Accelerometer WGT3X-BT, from which we can collect steps data. From this primary outcome measure we will also assess the change in number of steps taken comparing the first week to the following month after the intervention.
  Assuming mean enrollment number of steps per day is 9,302.29, we can detect an average increase of 2,500 steps per day with alpha set to 0.05 with 80% power.

SECONDARY OUTCOMES:
Time spent in moderate to vigorous physical activity | 5 weeks
  We will also analyze the time spent in moderate to vigorous physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: David Friedman, MD, MPH, PhD, Principal Investigator — Johns Hopkins University; Yuanbo Liang, MD, PhD, Principal Investigator — Clinical & Epidemiological Eye Research Centre, The affiliated eye hospital of Wenzhou Medical University
Locations (1):
- The affiliated eye hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China